CLINICAL TRIAL: NCT03506139
Title: Phase II Study of High Dose Radiotherapy and Concurrent Temozolomide Using Biologically-based Target Volume Definition in Patients With Newly Diagnosed Glioblastoma
Brief Title: Biologically-based Target Volumes to Treat Newly Diagnosed Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not funded
Sponsor: John M. Buatti (Other)
Collaborators: Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, John M. Buatti, Professor & Chair, Department of Radiation Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201801819
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
Keywords: Radiotherapy; Magnetic Resonance Imaging
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Intervention Model Description: Group treated to 75 Gray of radiation to at-risk target
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation Therapy (Experimental): External beam radiation therapy delivered to target volume.
  Interventions: Radiation: External beam radiation therapy

INTERVENTIONS:
Radiation: External beam radiation therapy — Radiotherapy to 75 Gy Radiation delivered 1 fraction / day, Monday through Friday, for a total of 30 fractions
  Other Names: radiotherapy; radiation

SUMMARY:
This clinical trial increases radiation to areas of the brain considered to be at risk for cancer. The at-risk areas are identified by a biological MRI scan. The study will look at side effects of the radiation and overall survival.

DETAILED DESCRIPTION:
This study evaluates if increasing radiation dose to at-risk areas impacts overall survival without causing a decrease in quality of life or an increase in radiation side effects.

Standard radiation dose for glioblastoma (GBM) is 60 Gray in 30 fractions, with patients receiving 1 fraction per day, Monday through Friday.

This trial will use a total of 75 Gray in 30 fractions, with participants receiving 1 fraction per day, Monday through Friday. Participants will still receive the standard chemotherapy (temozolomide) at the standard dose (75 mg/m2, once daily, 7 days a week).

This study also uses a different imaging technique to identify the tumor target and the tissues at risk. Normal imaging techniques will be used to define the standard target volume and will receive the standard radiation dose (60 Gray). A special MRI sequence will identify at risk areas based on diffusion and perfusion abnormalities. This area will receive the higher radiation dose (75 Gray).

Participants will also be asked to complete quality of life questionnaires and neurocognitive evaluations at specific time points. This is to identify any side effects from the higher radiation dose. Preliminary work done at University of Michigan suggests a lack of side effects from the higher dose of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to provide informed consent
* Newly diagnosed, histologically-confirmed supratentorial WHO grade IV gliomas including glioblastoma (all variants) and gliosarcoma.
* Patients must be 18 years of age or older.≥
* Karnofsky performance status ≥ 70
* Minimal life expectancy of 12 weeks.
* Maximal contiguous volume of tumor based on high b-value diffusion MRI and perfusion MRI < 1/3 volume of brain
* Patients must be treated within 6 weeks of most recent resection

Within 21 days of radiation fraction 1, the following blood test parameters must be met:

* Hemoglobin ≥ 10 g/dL (transfusion is acceptable)
* absolute neutrophils ≥ 1500/mm3
* platelet count ≥ 100,000/mm3
* total bilirubin ≤ 2 x upper limit of normal (ULN) (unless elevated bilirubin is related to Gilbert syndrome)
* ALT and AST ≤ 5 x ULN
* serum creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Recurrent glioma, or tumor involving the brainstem or cerebellum. Prior low-grade glioma without prior RT, now with malignant progression are eligible.
* Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment is not permitted. Prior chemotherapy for a different cancer is allowable if interval since last treatment cycle completion is >3 years.
* Evidence of CSF dissemination (positive CSF cytology for malignancy or MRI findings consistent with CSF dissemination).
* Multifocal disease (>1 lobe of involvement) of discontiguous, contrast enhancing disease as seen on conventional MRI
* Evidence of severe concurrent disease requiring treatment
* Known active malignancy as determined by treating medical and radiation oncologist
* Patients unable to undergo MRI exams
* Patients treated with previous cranial or head/neck radiotherapy leading to significant radiation field overlap.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring inpatient hospitalization or delay treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or compromise subject safety.
* Pregnant women are excluded from this study because ionizing radiation is a known teratogen, and temozolomide is a Class D agent with the potential for teratogenic or abortifacient effects.
* Nursing mothers declining to discontinue breastfeeding are excluded because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temozolomide.
* Patients with reproductive potential declining to use an effective contraceptive method during treatment are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 months after completing radiation therapy
  Estimate 12-month overall survival of GBM patients treated with 75 Gray of radiation based on advanced MRI planning, with concurrent temozolomide.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Every 2 months, for up to 60 months after completing radiation therapy, until progression or death from any cause
  Estimate progression-free survival (PFS) in GBM patients treated with 75 Gray of radiation based on advanced MRI planning, with concurrent temozolomide.
Identifying tissue at risk of recurrence | 12 months after completing radiation therapy
  Assess the ability of pre-treatment and mid-treatment advanced MRI to determine areas at high risk of recurrence
Distinguish progression from pseudoprogression | 12 months after completing radiation therapy
  Assess the ability of post-treatment advanced MRI to distinguish progression from pseudoprogression
Adverse events related to treatment | Weekly during radiation therapy, every 2 months post-radiation therapy for 7 months, then 13 & 19 months post-radiation
  Provide descriptive data regarding health-related quality of life (QOL), symptoms and neurocognitive function

CONTACTS AND LOCATIONS:
Overall Officials: John M. Buatti, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Department of Radiation Oncology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Individual participant data will be shared with a signed usage agreement. Additionally, a contract will be required between University of Iowa and the receiving institution.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request
Access Criteria: Email study contacts with request

REFERENCES:
- [Background] Hamstra DA, Galban CJ, Meyer CR, Johnson TD, Sundgren PC, Tsien C, Lawrence TS, Junck L, Ross DJ, Rehemtulla A, Ross BD, Chenevert TL. Functional diffusion map as an early imaging biomarker for high-grade glioma: correlation with conventional radiologic response and overall survival. J Clin Oncol. 2008 Jul 10;26(20):3387-94. doi: 10.1200/JCO.2007.15.2363. Epub 2008 Jun 9. PMID 18541899
- [Background] Galban CJ, Chenevert TL, Meyer CR, Tsien C, Lawrence TS, Hamstra DA, Junck L, Sundgren PC, Johnson TD, Galban S, Sebolt-Leopold JS, Rehemtulla A, Ross BD. Prospective analysis of parametric response map-derived MRI biomarkers: identification of early and distinct glioma response patterns not predicted by standard radiographic assessment. Clin Cancer Res. 2011 Jul 15;17(14):4751-60. doi: 10.1158/1078-0432.CCR-10-2098. Epub 2011 Apr 28. PMID 21527563